CLINICAL TRIAL: NCT07216456
Title: Improving Engagement With Vaginal Dilator Therapy After Pelvic Radiation: A Pilot Randomized Controlled Trial
Brief Title: Vaginal Dilator Therapy After Pelvic Radiation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00118002; 1K08CA304375 (NIH)
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Pelvic Radiotherapy; Vaginal Stenosis; Pelvic Cancer; Gynecologic Cancers; Anorectal Cancer; Urologic Cancer
Keywords: vaginal dilator therapy; pelvic radiation
MeSH Terms: conditions — Pelvic Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improving Engagement with Vaginal Dilator Therapy after Pelvic Radiation (Experimental): A 6-session (45 minutes each) behavioral intervention will be delivered individually and remotely via videoconferencing. The intervention will be designed to improve engagement with vaginal dilator therapy among female cancer survivors who underwent pelvic radiation therapy. The intervention includes coping strategies from cognitive behavioral therapy (e.g., progressive muscle relaxation) and acceptance and commitment therapy (e.g., mindfulness), as well as psychoeducation (e.g., how to use dilators), to enhance engagement with vaginal dilator therapy.
  Interventions: Behavioral: Improving Engagement with Vaginal Dilator Therapy after Pelvic Radiation
- Enhanced Usual Care (No Intervention): Written materials will highlight the purpose of dilator therapy and how to use dilators (including frequency and duration).

INTERVENTIONS:
Behavioral: Improving Engagement with Vaginal Dilator Therapy after Pelvic Radiation — The intervention includes coping strategies from cognitive behavioral therapy (e.g., progressive muscle relaxation) and acceptance and commitment therapy (e.g., mindfulness), as well as psychoeducation (e.g., how to use dilators), to enhance engagement with vaginal dilator therapy.
  Arms: Improving Engagement with Vaginal Dilator Therapy after Pelvic Radiation

SUMMARY:
This study is testing a new program to help women who have had pelvic radiation therapy to use vaginal dilators more regularly. Vaginal dilators are important tools that can help prevent or treat vaginal narrowing (called vaginal stenosis), which can happen after radiation and make medical exams or sexual activity painful or difficult. Even though dilators are recommended, many women don't use them as often as needed.

In this study, 88 participants will be randomly assigned to one of two groups:

* One group will receive the new behavioral program, which includes support and strategies to help with regular dilator use.
* The other group will receive written educational materials (enhanced usual care).

The study will look at how often and how long participants use their dilators, and whether the program helps reduce symptoms like pain or emotional distress. Participants will complete surveys at the beginning of the study and again at 3, 6, and 9 months, plus short monthly check-ins.

The goal is to see if the program is helpful and easy to use, and to prepare for a larger study in the future.

DETAILED DESCRIPTION:
This study is testing a new behavioral program to help women who have had pelvic radiation therapy use vaginal dilators more regularly. Vaginal dilators are important tools that help prevent or treat vaginal stenosis-a condition where the vagina becomes shorter or narrower after radiation. This can make medical exams and sexual activity painful or difficult. Although dilators are commonly recommended, many women struggle to use them consistently.

The new program is designed to support women in overcoming common challenges to using dilators, such as pain, emotional distress, and lack of information. It includes strategies from cognitive behavioral therapy and acceptance and commitment therapy, and is based on the Health Belief Model, which helps people understand how their beliefs affect their health behaviors.

The study will include 88 participants who will be randomly assigned to one of two groups:

* One group will receive the new behavioral program.
* The other group will receive written educational materials (enhanced usual care).

Participants will complete surveys at the beginning of the study and again at 3, 6, and 9 months. They will also complete short monthly check-ins to report how often and how long they use their dilators.

The main goals of the study are to:

* See if the program is easy to use and acceptable to participants.
* Track how often participants use their dilators.
* Measure changes in symptoms, emotional distress, and knowledge about dilator therapy.

This pilot study will help researchers prepare for a larger study in the future and improve support for women recovering from pelvic radiation.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* adults aged 18 years or older
* diagnosed with cancer of the anus, anal canal, anorectum, cervix, uterus, vagina, vulva, and/or bladder
* completed pelvic radiation therapy in the past year
* dilator therapy recommended by medical provider and standardized dilator received from provider
* able to speak/read English

Exclusion Criteria:

* aged less than 17 years
* under the care of a pelvic floor physical therapist at the time of study enrollment
* have a major/serious psychiatric concern (e.g., schizophrenia) as indicated by medical chart/medical provider
* inability to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2027-08-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility, as Measured by Session Completion and Attrition | 3 months post-baseline
  Feasibility will be determined by 1) greater than or equal to 80% of sessions completed and 2) attrition rate of less than or equal to 20%.
Acceptability, as Measured by the Treatment Acceptability Questionnaire | 3 months post-baseline
  Acceptability will be determined by average score of 5 or greater on the Treatment Acceptability Questionnaire (TAQ). The TAQ is a six-item measure assessing perceptions of an interventions acceptability, ethics, and effectiveness. Items are rated on a 7-point Likert scale, from "very unacceptable" to "very acceptable".

SECONDARY OUTCOMES:
Change in Dilator Therapy Use | From baseline to end of study enrollment at 9 months
  Dilator therapy use will be assessed monthly via text survey by four items used in prior research to assess average frequency of dilator use, average duration of dilator use per dilation, frequency of penetrative sexual activity, and frequency of alternate dilator use over the past month.
Completion of cancer screening | From baseline to end of study enrollment at 9 months
  Completion of cancer screening/surveillance that involved a pelvic exam will be assessed by asking one item about the frequency of completing recommended pelvic exams for cancer screening/surveillance in the past three months. This will be assessed every 3 months via self-report.
Change in symptoms, as measured by the Edmonton Symptom Assessment System | From baseline to end of study enrollment at 9 months
  The Edmonton Symptom Assessment System is a 10-item self-report scale of 9 common symptoms experienced by cancer patients. There is a 10th item in which patients can write in and rate another specific symptom experienced. Participants are asked to rate individual symptom burden on an 11 point scale (0-10) with higher scores indicating greater symptom burden. This will be assessed every 3 months by self-report.
Change in depressive symptoms, as measured by the PROMIS Depression Short Form | From baseline to end of study enrollment at 9 months
  Depressive symptoms will be assessed using the PROMIS Depression Short Form. This is an 8-item measure assessing symptoms of depression experienced over the last week. Participants will be asked to respond to items (e.g., "I felt sad," "I felt helpless") using a five-point scale ranging from "1" (never) to "5" (always). This will be assessed every 3 months by self-report.
Change in psychological flexibility, as measured by the Acceptance and Action Questionnaire II | From baseline to end of study enrollment at 9 months
  The Acceptance and Action Questionnaire II (AAQ-II) is a 7-item measure of psychological flexibility. Participants are asked to rate items on a 7-point scale from "1" (never true) to "7" (always true) and item scores are summed to create a total score between 7 and 49. Higher scores indicate lower psychological flexibility. This will be assessed every 3 months by self-report.
Change in understanding of psychosocial changes as measured by the modified Knowledge Scale | From baseline to end of study enrollment at 9 months
  A 14-item modified version of a Knowledge Scale developed by previous researchers will be used to assess understanding of psychosexual changes following pelvic radiation therapy and use and purpose of vaginal dilator therapy and other rehabilitation strategies. Higher summed scores on the knowledge scale indicate greater knowledge. This will be assessed every 3 months by self-report.
Change in self-efficacy, as measured by the modified Generalized Self-Efficacy Scale | From baseline to end of study enrollment at 9 months
  The Generalized Self-Efficacy Scale is a 10-item measure of self-efficacy. Respondents are asked to rate individuals items on a 4 point scale from "1" (not at all true) to "4" (exactly true). Items on this measure will be modified to assess self-efficacy with engaging in dilator therapy. Scores will be summed for a total between 10 and 40. Higher summed scores indicate greater self-efficacy to engage in dilator therapy. This will be assessed every 3 months by self-report.
Change in perceived susceptibility to developing vaginal stenosis, benefits and barriers to engaging in dilator therapy, as measured by the modified susceptibility, Benefits and Barriers Scale | From baseline to end of study enrollment at 9 months
  The 19-item Revised Susceptibility, Benefits, and Barriers Scale for mammography screening will be modified to assess perceived susceptibility to developing vaginal stenosis, benefits to engaging in dilator therapy, and barriers to engaging in dilator therapy. Items are rated on a 5-point Likert-type scale from "1" (strongly agree) to "5" (strongly disagree). Higher subscale scores indicate a lower degree of perceived susceptibility, benefits, and barriers, respectively. This will be assessed every 3 months by self-report.
Change in cues that prompt health-promoting behaviors, as measured by the modified Cues to Health Action Questionnaire | From baseline to end of study enrollment at 9 months
  The Cues to Health Action Questionnaire is a 32-item measure assessing cues that prompt health-promoting behaviors. The specific target action that will be emphasized in measure instructions is engaging in dilator therapy. Respondents will be asked to rank order specific cues to action for engaging dilator therapy. This will be assessed every 3 months by self-report.
Change in sexual feelings and responses, as measured by the Female Sexual Function Index | From baseline to end of study enrollment at 9 months
  The Female Sexual Function Index (FSFI) is a 19-item measure assessing sexual feelings and responses over the past 4 weeks. Participants are asked to rate individual items on a 5 or 6 point Likert-type scales, ranging from "0" or "1" to "5", with higher total score indicating greater sexual functioning. This will be assessed every 3 months by self-report.
Change in anxiety symptoms, as measured by the PROMIS Anxiety Short-Form | From baseline to end of study enrollment at 9 months
  The PROMIS Anxiety Short Form will be used to assess anxiety symptoms. This is an 7-item measure assessing symptoms of anxiety experienced over the last week. Participants will be asked to respond to items using a five-point scale ranging from "1" (never) to "5" (always). Responses will be summed for a total score between 7 and 35, with higher scores indicating higher levels of anxiety symptoms. This will be assessed every 3 months by self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Juliann Stalls, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
It is our intention to make all data generated from this proposal freely available after it is de-identified. Respondent identifiers will not be shared. All other scientific data (scale composites) will be both preserved and shared. The following data will be preserved and shared: qualitative data, patient-reported data from study assessments, and sociodemographic and medical data collected via patient report and health record. Researchers will make every effort to provide raw data in a non-proprietary format wherever possible to enhance reproducibility.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared either at the time of publication or at the end of the performance period, whichever comes first. All data deposited with the Duke Research Data Repository will be retained for a minimum of 25 years according to their stated Retention Policy.